CLINICAL TRIAL: NCT03980353
Title: Evaluation of Difficulties and Obstacles to the Integration in Community of Children With Type 1 Diabetes Before Primary School, Followed by the Diabetology Department of Lyon Pediatric Hospital.
Brief Title: Difficulties and Obstacles to the Integration in Community of Children With Type 1 Diabetes Before Primary School.
Acronym: DIABECO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0218; 2019-A01571-56 (Other: ID-RCB)
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children before entrance in primary school: Children with type 1 diabetes, who are too young to go to primary school at the start of the school year 2018-2019, followed in the Diabetology Department of Lyon Pediatric Hospital.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — The questionnaires have two parts: a general part and a second part focused on the integration in community of the type 1 diabetes children with specific questions about blood glucose, mealtimes, sporting activities and school trips.

SUMMARY:
The incidence of type 1 diabetes is increasing worldwide and in France, including among young children.

Type 1 diabetes has consequences for integration in community, especially on the management of hypoglycemia and hyperglycemia, mealtimes, participation in sporting activities and school trips.

This works' purpose is to describe obstacles and difficulties to the integration in community before primary school (day care center, childminder, and nursery school) of a complete sample of children with type 1 diabetes followed in the Diabetology Department of Lyon Pediatric Hospital, at the start of the school year 2018-2019. The investigating team will carry out a descriptive study, using different questionnaires addressed to the professionals (nursery school directors, day care nursery directors, childminders, school doctors, pediatricians and doctors of child and maternal protection centers) and to the parents of children with type 1 diabetes. These different questionnaires will help to take into account different points of view, in order to identify all the obstacles to integration of children with type 1 diabetes in community.

Through this work, secondary information actions through training and/or information leaflets will be carried out in order to facilitate the reception of these children in the community.

ELIGIBILITY:
Inclusion Criteria:

Children:

* Type 1 Diabetes
* Followed in the diabetology department of Lyon pediatric hospital
* Who are too young to go to primary school in 2018-2019
* Residing in the Rhône-Alpes region of France
* No parental opposition to the completion of the questionnaire (reflection period of 15 days after receipt the leaflet information)

For school directors, school doctors, pediatricians, child and maternal protection center doctors

* Questionnaire responses will be considered as evidence of no opposition.

Directors of nurseries and childminders who will agree to answer the telephone questionnaire after parents allow the study team to contact them

Exclusion Criteria:

Children:

* Child requiring another facilities for school (food allergies, celiac disease…)
* Language barrier not permitting a response to the questionnaires

For childminders and nursery directors

* refusal of parents to contact them
* refusal to participate declared during the telephone interview

For school directors, doctors and school doctors

* No prior involvement in the reception in community of a type 1 diabetes child

Ages: 12 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 1 year to 8 years old with Type 1 diabetes followed by the Diabetology Department of Lyon Pediatric Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Identification of community integration obstacles for children with type 1 diabetes | 15 minutes
  Participants will respond to a multi-question interview by telephone or a paper questionnaire. The questions will focus on the child's lifestyle (such as meal times, activities, blood glucose levels...) in order to identify integration obstacles

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie BENDELAC, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Service d'endocrinologie pédiatrique Hôpital Femme mère enfant, Bron, France